CLINICAL TRIAL: NCT04278404
Title: Pharmacokinetics, Pharmacodynamics, and Safety Profile of Understudied Drugs
Brief Title: Pharmacokinetics, Pharmacodynamics, and Safety Profile of Understudied Drugs Administered to Children Per Standard of Care (POPS)
Acronym: POPS or POP02
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Emmes Company, LLC (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00103838
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Coronavirus Infection (COVID-19); Pulmonary Arterial Hypertension; Urinary Tract Infections in Children; Hypertension; Pain; Hyperphosphatemia; Primary Hyperaldosteronism; Edema; Hypokalemia; Heart Failure; Hemophilia; Menorrhagia; Insomnia; Pneumonia; Skin Infection; Arrythmia; Asthma in Children; Bronchopulmonary Dysplasia; Adrenal Insufficiency; Fibrinolysis; Hemorrhage; Attention Deficit Hyperactivity Disorder; Multisystem Inflammatory Syndrome in Children (MIS-C); Kawasaki Disease; Coagulation Disorder; Down Syndrome
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pulmonary Arterial Hypertension; Hypertension; Pain; Hyperphosphatemia; Hyperaldosteronism; Edema; Hypokalemia; Heart Failure; Hemophilia A; Menorrhagia; Sleep Initiation and Maintenance Disorders; Pneumonia; Cellulitis; Arrhythmias, Cardiac; Bronchopulmonary Dysplasia; Adrenal Insufficiency; Hemorrhage; Attention Deficit Disorder with Hyperactivity; pediatric multisystem inflammatory disease, COVID-19 related; Mucocutaneous Lymph Node Syndrome; Hemostatic Disorders; Down Syndrome | interventions — Aminocaproic Acid; Amiodarone; Bosentan; Budesonide; Cefdinir; Cefepime; Ceftazidime; Clindamycin; Clobazam; Dexamethasone; Dexmedetomidine; SLI381; Fosfomycin; Furosemide; Gabapentin; Guanfacine; Hydrocortisone; Labetalol; Meropenem; Metformin; Milrinone; Nalbuphine; Nicardipine; Nifedipine; Oseltamivir; Oxycodone; Risperidone; Sertraline; Sevelamer; Spironolactone; Terbutaline; Tranexamic Acid; Voriconazole; Zolpidem; Azithromycin; Lopinavir; Ribavirin; tocilizumab; Interleukin 1 Receptor Antagonist Protein; Aspirin; canakinumab; Colchicine; Interferons; remdesivir; ruxolitinib; sarilumab; Abatacept; Infliximab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, effluent samples, and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and young adults who are prescribed drugs of interest: Children and young adults who are prescribed drugs of interest as part of their routine medical care OR are SARS-CoV-2 positive.
  Interventions: Drug: The POP02 study is collecting bodily fluid samples (i.e., whole blood, effluent samples) of children prescribed the following drugs of interest per standard of care:

INTERVENTIONS:
Drug: The POP02 study is collecting bodily fluid samples (i.e., whole blood, effluent samples) of children prescribed the following drugs of interest per standard of care: — The prescribing of drugs to children is not part of this protocol. Participants will receive DOIs as prescribed by their treating provider.
  Other Names: Aminocaproic acid; Amiodarone; Bosentan; Budesonide; Cefdinir; Cefepime; Ceftazidime; Clindamycin; Clobazam; Dexamethasone; Dexmedetomidine; Dextroamphetamine/Amphetamine; Fosfomycin; Furosemide; Gabapentin; Guanfacine; Hydrocortisone; Labetalol; Meropenem; Metformin; Milrinone; Nalbuphine; Nicardipine; Nifedipine; Oseltamivir; Oxycodone; Risperidone; Sertraline; Sevelamer Carbonate / Sevelamer Hydrochloride; Spironolactone; Terbutaline; Tranexamic acid; Voriconazole; Zolpidem; Azithromycin; Lopinavir/Ritonavir; Ribavirin; Tocilizumab; Anakinra; Aspirin; Canakinumab; Colchicine; Interferon; Remdesivir; Ruxolitinib; Sarilumab; Abatacept; Infliximab

SUMMARY:
The study investigators are interested in learning more about how drugs, that are given to children by their health care provider, act in the bodies of children and young adults in hopes to find the most safe and effective dose for children. The primary objective of this study is to evaluate the PK of understudied drugs currently being administered to children per SOC as prescribed by their treating provider.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is < 21 years of age
2. Parent/ Legal Guardian/ Adult Participant can understand the consent process and is willing to provide informed consent/HIPAA:
3. (a) Participant is receiving one or more of the study drugs of interest at the time of enrollment or (b) Participant is NOT receiving one or more of the study drugs of interest but is SARS-COV-2 positive within 60 days prior to enrollment

Exclusion Criteria:

1. Participant has a known pregnancy

   Below exclusion criteria apply only to:

   Participants receiving one or more of the study drugs of interest at the time of enrollment, DOI administration or PK sampling: (Refer to DOI specific appendices for details on enrollment cohort specifications and additional eligibility criteria)
2. Has had intermittent dialysis within previous 24 hours
3. Has had a kidney transplant within previous 30 days
4. Has had a liver transplant within previous 1 year
5. Has had a stem cell transplant within previous 1 year
6. Has had therapeutic hypothermia within previous 24 hours
7. Has had plasmapheresis within the previous 24 hours
8. Has a Ventricular Assist Device
9. Has any condition which would make the participant, in the opinion of the investigator, unsuitable for the study

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children under 21 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Clearance (CL) or apparent oral clearance (CL/F) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.
Volume of distribution (V) or apparent oral volume of distribution (V/F) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.
Elimination rate constant (ke) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.
Half-life (t1/2) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.
Absorption rate constant (ka) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.
AUC (area under the curve) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.
Maximum concentration (Cmax) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.
Time to achieve maximum concentration (Tmax) as measured by PK sampling | Data will be collected up to 90 days from the time of consent. For participants with Down Syndrome enrolling at sites designated as Down Syndrome sites, participants will be in the study for up to 210 days.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hornik, Principal Investigator — Duke Clinical Research Institute
Locations (49):
- United States (47):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Colorado University Denver, Aurora, Colorado
  - The Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - University of Florida Jacksonville Shands Medical Center, Jacksonville, Florida
  - Kapiolani Womens and Childrens Medical Center, Honolulu, Hawaii
  - Ann and Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - University of Kansas Medical Center-JG Kidney Institute, Kansas City, Kansas
  - University of Louisville Norton Childrens Hospital, Louisville, Kentucky
  - Tulane University Health Science Center, New Orleans, Louisiana
  - Ochsner Baptist Clinical Trials Unit, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Lexington, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Board of Regents of the University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Pennsylvania State University--Hershey Children's Hospital, Hershey, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina
  - Avera McKennan Hospital & University Medical Center, Sioux Falls, South Dakota
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas-Southwestern Medical Center Dallas, Dallas, Texas
  - University of Texas--Memorial Hermann Texas Medical Center, Houston, Texas
  - The Womens Hospital of Texas, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - University Wisconsin Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tremoulet A, Le J, Poindexter B, Sullivan JE, Laughon M, Delmore P, Salgado A, Ian-U Chong S, Melloni C, Gao J, Benjamin DK Jr, Capparelli EV, Cohen-Wolkowiez M; Administrative Core Committee of the Best Pharmaceuticals for Children Act-Pediatric Trials Network. Characterization of the population pharmacokinetics of ampicillin in neonates using an opportunistic study design. Antimicrob Agents Chemother. 2014 Jun;58(6):3013-20. doi: 10.1128/AAC.02374-13. Epub 2014 Mar 10. PMID 24614374
- [Background] Hornik CP, Benjamin DK Jr, Smith PB, Pencina MJ, Tremoulet AH, Capparelli EV, Ericson JE, Clark RH, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act-Pediatric Trials Network. Electronic Health Records and Pharmacokinetic Modeling to Assess the Relationship between Ampicillin Exposure and Seizure Risk in Neonates. J Pediatr. 2016 Nov;178:125-129.e1. doi: 10.1016/j.jpeds.2016.07.011. Epub 2016 Aug 10. PMID 27522443
- [Background] Le J, Poindexter B, Sullivan JE, Laughon M, Delmore P, Blackford M, Yogev R, James LP, Melloni C, Harper B, Mitchell J, Benjamin DK Jr, Boakye-Agyeman F, Cohen-Wolkowiez M. Comparative Analysis of Ampicillin Plasma and Dried Blood Spot Pharmacokinetics in Neonates. Ther Drug Monit. 2018 Feb;40(1):103-108. doi: 10.1097/FTD.0000000000000466. PMID 29271816
- [Background] Gonzalez D, Melloni C, Yogev R, Poindexter BB, Mendley SR, Delmore P, Sullivan JE, Autmizguine J, Lewandowski A, Harper B, Watt KM, Lewis KC, Capparelli EV, Benjamin DK Jr, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act - Pediatric Trials Network Administrative Core Committee. Use of opportunistic clinical data and a population pharmacokinetic model to support dosing of clindamycin for premature infants to adolescents. Clin Pharmacol Ther. 2014 Oct;96(4):429-37. doi: 10.1038/clpt.2014.134. Epub 2014 Jun 20. PMID 24949994
- [Background] Gonzalez D, Delmore P, Bloom BT, Cotten CM, Poindexter BB, McGowan E, Shattuck K, Bradford KK, Smith PB, Cohen-Wolkowiez M, Morris M, Yin W, Benjamin DK Jr, Laughon MM. Clindamycin Pharmacokinetics and Safety in Preterm and Term Infants. Antimicrob Agents Chemother. 2016 Apr 22;60(5):2888-94. doi: 10.1128/AAC.03086-15. Print 2016 May. PMID 26926644
- [Background] Gonzalez D, Melloni C, Poindexter BB, Yogev R, Atz AM, Sullivan JE, Mendley SR, Delmore P, Delinsky A, Zimmerman K, Lewandowski A, Harper B, Lewis KC, Benjamin DK Jr, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act--Pediatric Trials Network Administrative Core Committee. Simultaneous determination of trimethoprim and sulfamethoxazole in dried plasma and urine spots. Bioanalysis. 2015;7(9):1137-49. doi: 10.4155/bio.15.38. PMID 26039810
- [Background] Autmizguine J, Melloni C, Hornik CP, Dallefeld S, Harper B, Yogev R, Sullivan JE, Atz AM, Al-Uzri A, Mendley S, Poindexter B, Mitchell J, Lewandowski A, Delmore P, Cohen-Wolkowiez M, Gonzalez D; the Pediatric Trials Network Steering Committee. Population Pharmacokinetics of Trimethoprim-Sulfamethoxazole in Infants and Children. Antimicrob Agents Chemother. 2017 Dec 21;62(1):e01813-17. doi: 10.1128/AAC.01813-17. Print 2018 Jan. PMID 29084742
- [Background] Dallefeld SH, Atz AM, Yogev R, Sullivan JE, Al-Uzri A, Mendley SR, Laughon M, Hornik CP, Melloni C, Harper B, Lewandowski A, Mitchell J, Wu H, Green TP, Cohen-Wolkowiez M. A pharmacokinetic model for amiodarone in infants developed from an opportunistic sampling trial and published literature data. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):419-430. doi: 10.1007/s10928-018-9576-y. Epub 2018 Feb 12. PMID 29435949
- [Background] Hornik CP, Gonzalez D, van den Anker J, Atz AM, Yogev R, Poindexter BB, Ng KC, Delmore P, Harper BL, Melloni C, Lewandowski A, Gelber C, Cohen-Wolkowiez M, Lee JH; Pediatric Trial Network Steering Committee. Population Pharmacokinetics of Intramuscular and Intravenous Ketamine in Children. J Clin Pharmacol. 2018 Aug;58(8):1092-1104. doi: 10.1002/jcph.1116. Epub 2018 Apr 20. PMID 29677389
- [Background] Drolet BA, Boakye-Agyeman F, Harper B, Holland K, Lewandowski A, Stefanko N, Melloni C; Pediatric Trials Network Steering Committee (See Acknowledgments for a listing of committee members.). Systemic timolol exposure following topical application to infantile hemangiomas. J Am Acad Dermatol. 2020 Mar;82(3):733-736. doi: 10.1016/j.jaad.2019.02.029. Epub 2019 Feb 18. No abstract available. PMID 30790601
- [Background] Hornik CP, Yogev R, Mourani PM, Watt KM, Sullivan JE, Atz AM, Speicher D, Al-Uzri A, Adu-Darko M, Payne EH, Gelber CE, Lin S, Harper B, Melloni C, Cohen-Wolkowiez M, Gonzalez D; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Population Pharmacokinetics of Milrinone in Infants, Children, and Adolescents. J Clin Pharmacol. 2019 Dec;59(12):1606-1619. doi: 10.1002/jcph.1499. Epub 2019 Jul 17. PMID 31317556
- See also: Food and Drug Administration. General Clinical Pharmacology Considerations for Pediatric Studies for Drugs and Biological Products — http://www.fda.gov/media/90358/download
- See also: Extracorporeal Life Support Organization (ELSO). ECLS Registry Report: International Summary Ann Arbor, MI: Extracorporeal Life Support Organization (ELSO); 2020 — https://www.elso.org/Registry/Statistics/InternationalSummary.aspx
- See also: Wildschut E, editor. Drug therapies in neonates and children during extracorporeal membrane oxygenation (ECMO); Keep your eyes open. Rotterdam, The Netherlands: Erasmus MC; 2010. — https://pdfs.semanticscholar.org/b0d9/11f1f38ad7a83694bbee99fd41ae3db5b07d.pdf